CLINICAL TRIAL: NCT05966623
Title: Assessing the Impact of Vidéo Remote Sign Language Interpreting in Healthcare: Linking Disability Studies With Empirical Challenges of Public Health Research
Brief Title: Assessing the Impact of Vidéo Remote Sign Language Interpreting in Healthcare
Acronym: Impact of VRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: Universidad del Rosario (Other); Hospital Universitario Mayor Mederi (Unknown); Clinica Nuestra Senora de la Paz (Unknown)
Responsible Party: Principal Investigator, Minerva Rivas Velarde, Group Leader, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: -2021-05-50-M1
Record Dates: First submitted 2023-07-17; First posted 2023-07-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Intervention Model Description: Arm Intervention Experimental VRI sign language interpretation Participants will be welcome from their entry point to the hospital, they will attend a general check-up with a GP or other services and be provided with VRI until they leave Participants will be provided with a Tablet of 14' inches with interrupted VRI in Colombian Sign Language. Professionally accredited Sign language interpreter. At the end of the hospital visit, they will complete a scale measuring Doctor-Patient-Communication
  Experimental: primo control Participants get welcome at the entry point of the hospital, they will attend a general check-up with a GP or other services and they are not provided with by the study with VRI Participants get welcome at the entry point of the hospital, they are not provided with VRI. At the end of the hospital visit, they will complete a scale measuring Doctor-Patient-communication
Masking Description: Single-blinded - The researcher needs to learn before the patient comes to the hospital as VRI needs to be organised. Thus, they will only know if the participants shall be assigned to the intervention or control group after the patient agrees to take part. Double blinding is not feasible as interpreters will not be available 24x7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental VRI sign language interpretation (Experimental): Participants will be provided with a Tablet of 14' inches with interrupted VRI in Colombian Sign Language. Professionally accredited Sign language interpreter. At the end of the hospital visit, they will complete a scale measuring Doctor-Patient-Communication
  Interventions: Other: Video Remote Interpretation
- Experimental: primo control (No Intervention): Participants get welcome at the entry point of the hospital, they are not provided with VRI. At the end of the hospital visit, they will complete a scale measuring Doctor-Patient-communication

INTERVENTIONS:
Other: Video Remote Interpretation — To assess the effectiveness of the VRI system in improving communication outcomes between Deaf patients and doctors Produce a VRI model addressing the challenges faced by Deaf people that will be tested, implemented, and sustained in Bogota Colombia.
  Arms: Experimental VRI sign language interpretation

SUMMARY:
This is a randomise study that looks at what is the effectiveness of the VRI system in improving communication outcomes between Deaf patients and doctors versus the 'available standard of care of the usual communication tools, including informal interpretation, lip or note reading, using their mobile phones to contact a formal or informal interpreter, for Deaf patients aged 18 and older in Bogota Colombia

DETAILED DESCRIPTION:
Background and Rationale:

In-person or VRI sign language interpretation is largely unavailable. In a scoping review, the researchers identified a knowledge gap regarding the quality of interpretation and training in sign language interpretation for health care. The researchers also found that this area is under-researched, and the evidence is scant. All available evidence came from high-income countries, which is particularly problematic given that most DHH persons live in low- and middle-income countries. Thus, the available literature shows that VRI may enable deaf users to overcome interpretation barriers and can potentially improve communication outcomes between them and health personnel within health care services. For VRI to be acceptable, sign language users require a VRI system supported by devices with large screens and a reliable internet connection, as well as qualified interpreters trained in medical interpretation. There is no clear data on the availability of VRI or in-person interpretation. Given the cost, VRI may be more available than in person. Available data tend to focus on assessing personal references of Deaf users in regards to interpretation, as well as interpreters' preferences and maximising recourses allocation.

Objective(S):

To assess the effectiveness of the VRI system in improving communication outcomes between Deaf patients and doctors Produce a VRI model addressing the challenges faced by Deaf people that will be tested, implemented, and sustained in Bogota, Colombia.

Explanation for choice of comparator

In-person or VRI sign language interpretation is largely unavailable. Thus, there is no clear data on the magnitude of the availability gap of VRI or in-person interpretation. In-person qualified sign language interpretation in the healthcare setting tends to be described as the ideal standard of service provision. Thus, it is largely unavailable even in HIC. The assumption is based upon minimal available evidence on the personal preferences of Deaf persons in the USA. There is no evidence that in-person interpretation is efficient in the context of weaker infrastructure, such as low sign language literacy rates across Deaf persons, lack of standard qualification of interpreters and lack of interpreters and sustainable financing in HIC. To my knowledge, there is no study assessing DPC while using sign language interpretation.

Given the cost, VRI may be more sustainable than in-person. Assessing the efficiency of VRI versus the standard of care would be d of more value, given that there is no other effective intervention to compare.

ELIGIBILITY:
Inclusion Criteria:

* Uses Colombian Sign Language as the preferred language.
* Enough sensorimotor, cognitive and communication skills to communicate independently with health personnel

Exclusion Criteria:

* Does not communicate using sign language.
* Additional impairments which affect language development or the use of sign language.
* Refusal of the participant's representative(s) to participate in the study,
* Refusal of the participant's representative(s) to participate in a modality of the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Communication outcomes | 12 months
  The score of a selected' scale assesses A: creating a good interpersonal relationship, B: exchanging information, and C: Making treatment-related decisions that involve the patients in decision-making.
  The results of the scale will be asses using descriptive analytics (Fisher exact test will be applied to compare the 2 groups) Multiple regression analysis will be applied using demographic data and health indicators.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Clinica Nuestra Senora de la Paz, Bogotá
  - Hospital Universitario Mayor Mederi, Bogotá

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivas Velarde M, Izquierdo Martinez LC, Dalal J, Martinez-R A, Guevara Rojas KL, Parra Valero NA, Cruz Reyes DL, Cuculick J, Vallejo-Silva A, Irreno-Sotomonte J, Groce N. Video Remote Sign Language Interpreting and Health Communication for Deaf Patients: A Randomized Clinical Trial. JAMA Netw Open. 2026 Feb 2;9(2):e2557189. doi: 10.1001/jamanetworkopen.2025.57189. PMID 41637069
- [Derived] Rivas Velarde M, Izquierdo Martinez LC, Dalal J, Martinez-R A, Cruz Reyes DL, Cuculick J, Vallejo-Silva A, Irreno-Sotomonte J, Groce N. Video Remote Sign Language Interpreting in Health Communication for Deaf People: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 2;13:e64590. doi: 10.2196/64590. PMID 39622021